CLINICAL TRIAL: NCT04132037
Title: An Observational Study on Intermittent Self Catheterisation Discontinuation Factors in Multiple Sclerosis Patients
Acronym: SEPAS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Toulouse (Other)
Collaborators: French Association for Research on Multiple Sclerosis (Unknown)
Responsible Party: Sponsor
Other Study IDs: RC31/18/0354; 2019-A00327-50 (Other: ID-RCB)
Record Dates: First submitted 2019-10-09; First posted 2019-10-18 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Urinary disorders; Intermittent Self Catheterisation
MeSH Terms: conditions — Multiple Sclerosis | interventions — Electronic Health Records; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient with multiple sclerosis: At each visit, inclusion, 6 weeks, 6 months, 12 months, and 24 months, the clinical and urinary data will be recorded and the ISC frequency , ISC discontinuation and adherence scale will be evaluated
  Interventions: Other: data record

INTERVENTIONS:
Other: data record — At each protocol's visit, clinical and urinary data will be recorded and the answers of the questionnaires will be also reported
  Other Names: questionnaires

SUMMARY:
Urinary disorders (UD) are common in Multiple Sclerosis (MS) and can necessitate using Intermittent Self Catheterisation (ISC). It is well experienced by patients, has little impact on daily life and improves quality of life. However, studies are lacking on long-term adherence to this treatment as well as on discontinuation factors. Our main objective is to prospectively assessed factors associated with ISC discontinuation 2 years after having introduced this technique.

DETAILED DESCRIPTION:
Urinary disorders (UD) are common in Multiple Sclerosis (MS). About 65% of patients suffering from moderate to severe troubles. In case of voiding dysfunction, the reference treatment is based on intermittent self catheterisation (ISC). UD in spinal cord injury (SCI) patients have been widely studied. They are very common, and are life-threatening in the absence of appropriate care. Management of neurological UD (as those occurring in MS) are well defined. ISC is the gold standard of bladder emptying method in this pathological context, and has been the subject of numerous studies. In SCI, the ISC discontinuation rate varies from 52 to 80% according to the published studies, the main factors of continuation being the autonomy to perform the technique, and the continence rate. However, the results are variable. In case of MS, the studies are lacking, the results concerning the discontinuation rate and factors associated with discontinuation are poor. Our main objective within the French speaking neurology study group (GENULF), is to prospectively assessed factors associated with ISC discontinuation 2 years after having introduced this technique.

This predictive study will be multicenter, observational, analytical, and prospective and will not modify current clinical practice.

We will record clinical and urinary data at each visit (inclusion, 6 weeks, 6 months, 12 months, and 24 months). We will note also if the patient practice ISC as prescribed in order to identify discontinuation of the ISC.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 to 65 years
* Patient with MS
* First ISC prescription
* Patient giving informed consent
* Patient affiliated to the social security system

Exclusion Criteria:

* Patient who has already tried / practiced ISC
* Patient under safeguard of justice / guardianship / tutorship
* Pregnant or lactating woman

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple Sclerosis Patients requiring Intermittent Self Catheterisation
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2019-06-26 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
intermittent self catheterisation discontinuation at 2 years after the start of learning. | 2 years
  intermittent self catheterisation frequency and the adherence scorage will be evaluated for each patient.

SECONDARY OUTCOMES:
intermittent self catheterisation discontinuation at 6 weeks, after the start of learning. | 6 WEEKS
  intermittent self catheterisation frequency will be evaluated for each patient.
intermittent self catheterisation discontinuation 6 months after the start of learning. | 6 months
  intermittent self catheterisation frequency will be evaluated for each patient.
intermittent self catheterisation discontinuation at 1 year after the start of learning. | 1 year
  intermittent self catheterisation frequency will be evaluated for each patient.

CONTACTS AND LOCATIONS:
Overall Officials: castel lacanal EVELYNE, Principal Investigator — University Hospital, Toulouse
Locations (1):
- UHToulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No